CLINICAL TRIAL: NCT05583929
Title: an Investigation of the Relationship Between Walking Ability and Limit of Stability in Children With Spastic Cerebral Palsy
Brief Title: Walking Ability and Limit of Stability in Children With Spastic Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Bayram Sırrı, Phisical Therapist, Research Asistant, Master in Science, Muş Alparslan University
Other Study IDs: GO-22/398
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Gait, Spastic
Keywords: gait, walking ability, limit of stability, cerebral palsy
MeSH Terms: conditions — Gait Disorders, Neurologic; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spastic Cerebral Palsy: Children with spastic cerebral palsy
  Interventions: Other: GAITRite gaitway system, Bertec Balance System
- Healthy Developing Peers: Children with healthy developing peers
  Interventions: Other: GAITRite gaitway system, Bertec Balance System

INTERVENTIONS:
Other: GAITRite gaitway system, Bertec Balance System — GAITRite gaitway system will use to assess gait parameters, Bertec Balance System will use to assess limit of stability

SUMMARY:
Trunk control in children with spastic Cerebral Palsy (CP) is impaired. They have weaker trunk muscle strenght, and insufficient sitting/standing balance according to their developing peers. Since their weak trunk muscles and insufficient balance responses, they are not able to walk as functional similar to their peers. Additionaly limit of stability is worsen in children with CP. Investigation of the relationship between walking ability and limit of stability when seated position is important to understand which child is acceptable for training of walk. However we did not found any study to explain it. Therefore the aim of this study is to investigate walking ability and limit of stability in children with spastic CP, and to compare their developing peers.

ELIGIBILITY:
Inclusion Criteria:

* spastic serebral palsy, between the ages 6-15 years, between the I-IV. levels of GMFCS, be able to understand command given by physical therapist

Exclusion Criteria:

* undergone botulinum toxin A to upper and/or lower extremities, undergone any surgery to their extremities, be at the V. levels of GMFCS

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Spastic cerebral palsy and their developing peers
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Gait parameters (stride length in cm, step width in cm, time in swing phase in second, time in stance phase in second) | 20 minutes
  Gait parameters will be assessed by GAITRite walking way system.
Limit of stability when sitting and standing position in cm | 20 minutes
  Limit of stability will be evaluated by BERTEC balance system.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Sırrı, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided